CLINICAL TRIAL: NCT05512793
Title: PolyDeep Advance 2: Clinical Validation of PolyDeep. Randomized Clinical Trial with a Tandem Colonoscopy Design.
Brief Title: Clinical Validation of PolyDeep: an Artificial Intelligence-based Computer-aided Polyp Detection (CADe) and Characterization (CADx) System. Polydeep Advance 2.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government); Asociación Española de Gastroenterología (Other); Ministry of Work and Welfare - Xunta de Galicia (Other Government); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PolyDeep Advance 2.0
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Adenoma; Colorectal Serrated Lesions; Colorectal Polyps; Computer-Aided polyp Detection (CAD)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who fulfill criteria will be randomly allocated to perform the first withdrawal with the standard technique versus PolyDeep assisted colonoscopy. All colorectal detected polyps will be resected. After a second cecal intubation, second withdrawal will be performed with the opposite technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Technique followed by Combination (Active Comparator): Back-to-back tandem colonoscopies by the same endoscopist. The first colonoscopy will be performed without PolyDeep (standard technique) followed immediately by another colonoscopy with PolyDeep (combination technique).
  Interventions: Diagnostic Test: Standard technique First colonoscopy without PolyDeep
- Combination followed by Standard Technique (Active Comparator): Back-to-back tandem colonoscopies by the same endoscopist. In this arm, the first colonoscopy with be performed with PolyDeep (combination technique) followed immediately by another colonoscopy without PolyDeep (standard technique)
  Interventions: Diagnostic Test: Combination technique First colonoscopy with PolyDeep

INTERVENTIONS:
Diagnostic Test: Standard technique First colonoscopy without PolyDeep — Standard technique First colonoscopy without PolyDeep
  Arms: Standard Technique followed by Combination
Diagnostic Test: Combination technique First colonoscopy with PolyDeep — Combination technique First colonoscopy with PolyDeep
  Arms: Combination followed by Standard Technique

SUMMARY:
This study is a clinical validation of PolyDeep, a computer-aided polyp detection (CADe) and characterization (CADx) system. PolyDeep Advance 2 is a multicentric randomized clinical trial with a tandem colonoscopy design. The hypothesis of this study is that Polydeep assisted colonoscopy will reduce the number of missed adenomas in the first withdrawal.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the most frequently cancer in western world. A fundamental tool for detection and prevention is the colonoscopy. The detection and endoscopic resection of colorectal polyps, the precursor lesion of CRC, can reduce CRC incidence and mortality. Adenoma detection rate is the most used endoscopic quality indicator. The improvement of this indicator is related to the reduction of postcolonoscopy CRC incidence and mortality.

Colorectal polyp diagnosis is based on endoscopic resection and histological analysis. An accurate optical diagnosis could avoid histological lesion of smaller lesions, reducing the costs associated with histological diagnosis. The NICE (NBI International Colorectal Endoscopic) Classification has proposed the use of high definition endoscopes that have Narrow Band Imaging. However, NICE must be used by endoscopists who are sufficiently prepared and who have overcome the learning curve. Therefore, optical histology diagnosis with high accuracy independently of the center and the endoscopist is necessary.

Computer Aid Diagnosis (CAD) systems based on Artificial Intelligence are experiencing exponential development in the field of medical image analysis. The development of the CAD system is based on the creation of large databases of endoscopic images and/or videos, on the training, development and validation of diagnostic algorithms in such databases and, finally, on prospective clinical validation in patients undergoing colonoscopy. The goal of CAD systems in colonoscopy is double. First, it aims to increase the detection of polyps (CADe) in general, and of adenomas and serrated lesions in particular. The second objective is to characterize (CADx) the histology of detected lesion.

PolyDeep CAD is a functional prototype. It is capable of detecting, locating and classifying colorectal polyps. In vivo validation data shows that PolyDeep has high diagnostic accuracy for polyp identification and that this accuracy can be accommodated This clinical trial is part of the clinical validation of PolyDeep. We will perform a randomized clinical trial with a tandem colonoscopy design with adenoma miss rate as the main objective.

ELIGIBILITY:
Inclusion Criteria:

* First diagnostic colonoscopy performed after a positive fecal immunochemical test performed within the CRC screening program.
* Surveillance after colorectal adenomas resection.
* Authorization after reading the information sheet and singing the informed consent.

Exclusion Criteria:

* Incomplete colonoscopy without cecal intubation.
* Colonoscopies with insufficient intestinal cleansing (Boston Bowel Preparation Scale <6 or <2 in any of the evaluated segments).
* Detected lesions without histological diagnosis.
* Previous CRC.
* Previous colonic resection.
* CRC associated hereditary syndrome.
* Serrated polyposis syndrome.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Adenoma miss rate (AMR) | 1 Year
  AMR will be calculated as the number of adenomas detected on the withdrawal or portion in either group divided by the total number of adenomas detected during both withdrawals

SECONDARY OUTCOMES:
Polyp miss rate | 1 Year
  It will be calculated as the number of polyps detected on the withdrawal or portion in either group divided by the total number of polyps detected during both withdrawals
Serrated lesions miss rate | 1 Year
  It will be calculated as the number of serrated lesions detected on the withdrawal or portion in either group divided by the total number of serrated lesions detected during both withdrawals
Diagnostic yield and lesions characterization | 1 Year
  The diagnostic yield will be measure using sensitivity , specificity, Positive Predictive Value, Negative Predictive Value, likelihood ratios and Youden index. Histological diagnosis will be used as the gold standard.
Withdrawal time. (First/second colonoscopy) | 1 Year
  Withdrawal time between the two arms will be calculated and compared.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Complexo Hospitalario Universitario de Ourense, Ourense, Ourense
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra, Pontevedra
  - Hospital Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cubiella J, Marzo-Castillejo M, Mascort-Roca JJ, Amador-Romero FJ, Bellas-Beceiro B, Clofent-Vilaplana J, Carballal S, Ferrandiz-Santos J, Gimeno-Garcia AZ, Jover R, Mangas-Sanjuan C, Moreira L, Pellise M, Quintero E, Rodriguez-Camacho E, Vega-Villaamil P; Sociedad Espanola de Medicina de Familia y Comunitaria y Asociacion Espanola de Gastroenterologia. Clinical practice guideline. Diagnosis and prevention of colorectal cancer. 2018 Update. Gastroenterol Hepatol. 2018 Nov;41(9):585-596. doi: 10.1016/j.gastrohep.2018.07.012. Epub 2018 Sep 20. English, Spanish. PMID 30245076
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046
- [Background] ASGE Technology Committee; Abu Dayyeh BK, Thosani N, Konda V, Wallace MB, Rex DK, Chauhan SS, Hwang JH, Komanduri S, Manfredi M, Maple JT, Murad FM, Siddiqui UD, Banerjee S. ASGE Technology Committee systematic review and meta-analysis assessing the ASGE PIVI thresholds for adopting real-time endoscopic assessment of the histology of diminutive colorectal polyps. Gastrointest Endosc. 2015 Mar;81(3):502.e1-502.e16. doi: 10.1016/j.gie.2014.12.022. Epub 2015 Jan 16. PMID 25597420
- [Background] Puig I, Lopez-Ceron M, Arnau A, Rosinol O, Cuatrecasas M, Herreros-de-Tejada A, Ferrandez A, Serra-Burriel M, Nogales O, Vida F, de Castro L, Lopez-Vicente J, Vega P, Alvarez-Gonzalez MA, Gonzalez-Santiago J, Hernandez-Conde M, Diez-Redondo P, Rivero-Sanchez L, Gimeno-Garcia AZ, Burgos A, Garcia-Alonso FJ, Bustamante-Balen M, Martinez-Bauer E, Penas B, Pellise M; EndoCAR group, Spanish Gastroenterological Association and the Spanish Digestive Endoscopy Society. Accuracy of the Narrow-Band Imaging International Colorectal Endoscopic Classification System in Identification of Deep Invasion in Colorectal Polyps. Gastroenterology. 2019 Jan;156(1):75-87. doi: 10.1053/j.gastro.2018.10.004. Epub 2018 Oct 6. PMID 30296432
- [Background] Jin EH, Lee D, Bae JH, Kang HY, Kwak MS, Seo JY, Yang JI, Yang SY, Lim SH, Yim JY, Lim JH, Chung GE, Chung SJ, Choi JM, Han YM, Kang SJ, Lee J, Chan Kim H, Kim JS. Improved Accuracy in Optical Diagnosis of Colorectal Polyps Using Convolutional Neural Networks with Visual Explanations. Gastroenterology. 2020 Jun;158(8):2169-2179.e8. doi: 10.1053/j.gastro.2020.02.036. Epub 2020 Feb 29. PMID 32119927
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963
- [Background] Parmar R, Martel M, Rostom A, Barkun AN. Validated Scales for Colon Cleansing: A Systematic Review. Am J Gastroenterol. 2016 Feb;111(2):197-204; quiz 205. doi: 10.1038/ajg.2015.417. Epub 2016 Jan 19. PMID 26782820
- [Background] Parsa N, Rex DK, Byrne MF. Colorectal polyp characterization with standard endoscopy: Will Artificial Intelligence succeed where human eyes failed? Best Pract Res Clin Gastroenterol. 2021 Jun-Aug;52-53:101736. doi: 10.1016/j.bpg.2021.101736. Epub 2021 Feb 22. PMID 34172255
- [Background] Wani S, Rastogi A. Narrow-band imaging in the prediction of submucosal invasive colon cancer: how "NICE" is it? Gastrointest Endosc. 2013 Oct;78(4):633-6. doi: 10.1016/j.gie.2013.06.015. No abstract available. PMID 24054741
- [Background] Mangas-Sanjuan C, Santana E, Cubiella J, Rodriguez-Camacho E, Seoane A, Alvarez-Gonzalez MA, Suarez A, Alvarez-Garcia V, Gonzalez N, Lue A, Cid-Gomez L, Ponce M, Bujanda L, Portillo I, Pellise M, Diez-Redondo P, Herraiz M, Ono A, Pizarro A, Zapater P, Jover R; QUALISCOPIA Study Investigators. Variation in Colonoscopy Performance Measures According to Procedure Indication. Clin Gastroenterol Hepatol. 2020 May;18(5):1216-1223.e2. doi: 10.1016/j.cgh.2019.08.035. Epub 2019 Aug 22. PMID 31446179
- See also: Polydeep website — http://polydeep.org/
- See also: Effect of a deep-learning computer-aided detection system on adenoma detection during colonoscopy (CADe-DB trial): a double-blind randomised study. — https://linkinghub.elsevier.com/retrieve/pii/S246812531930411X